CLINICAL TRIAL: NCT04881578
Title: Atrial Fibrillation Before and After Patent Foramen Ovale Closure Study
Acronym: ALFA-ROMEO
Status: Active, not recruiting | Type: Observational
Sponsor: Raban Jeger (Other)
Responsible Party: Sponsor-Investigator, Raban Jeger, Prof. Dr. med., University Hospital, Basel, Switzerland
Organization: University Hospital, Basel, Switzerland (Other)
Other Study IDs: 2021-00016
Record Dates: First submitted 2021-05-05; First posted 2021-05-11 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Cryptogenic Stroke; Foramen Ovale, Patent; Atrial Fibrillation
Keywords: occlusion of patent foramen ovale
MeSH Terms: conditions — Ischemic Stroke; Foramen Ovale, Patent; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: continuous cardiac monitoring before and after transcatheter PFO closure — Data will be assessed from patients with cryptogenic stroke and planned PFO occlusion who undergo the contemporary ICM protocols to search for silent AF

SUMMARY:
The aim of the ALFA ROMEO study is to better understand the association between cryptogenic stroke, PFO, PFO closure and AF.

DETAILED DESCRIPTION:
For patients with cryptogenic stroke and PFO, a better understanding of the exact incidence of new-onset AF before and after PFO closure, its occurrence during follow-up, its persistence or reversibility and its prognostic impact is critical: If only a PFO, but no AF is available, then PFO closure followed by a limited duration of antiplatelet therapy is indicated. If on the other hand side a PFO and AF is found, lifelong therapeutic anticoagulation is mandatory.

By using the contemporary ICM protocols to search for silent AF in patients with cryptogenic stroke and a PFO for 3 months before PFO closure, ALFA ROMEO will help to understand the relationship of silent and previously undetected AF in the setting of PFO and investigate the true incidence of new-onset AF and its temporal course after effective PFO closure. Our findings will have the potential to impact on the future diagnostic and therapeutic management of patients with cryptogenic stroke and a PFO

ELIGIBILITY:
Inclusion Criteria:

1. History of embolic events such as cryptogenic stroke or systemic embolism (single event or multiple events). A stroke is considered to be cryptogenic if no possible cause can be determined despite extensive workup according to the standard protocol of the participating center (TOAST classification 5b) (29). Before inclusion in the study, the following tests are required as standard tests to establish the diagnosis of cryptogenic stroke:

   * MRI or computed tomography (CT) of the neurocranium (documenting ischemic embolic stroke)
   * 12-lead ECG (exclusion of AF)
   * Continuous ECG monitoring for at least 7 days (inpatient telemetry or Holter-ECG as an in- or outpatient
   * Ultrasonography, CT or MRI angiography of head and neck to rule out arterial disease as a cause of stroke (see below), or other potential causes of stroke
2. Cardiac monitoring is planned to be performed with the BIOMONITOR III(m) device
3. Presence of right-to-left shunt through a PFO as assessed by means of transesophageal echocardiography (TEE) with agitated saline while the patient is at rest or while a Valsalva maneuver is being performed.
4. Occlusion of PFO is planned to be performed with the AMPLATZERTM PFO OCCLUDER device.
5. Patient is willing to sign patient consent form.
6. Age ≥18 years.

Exclusion Criteria:

1. Known etiology of the embolic event (based on neuro-/cardiac/vascular imaging), such as:

   * Evidence of large-artery atherosclerosis (ultrasonography, CT or MRI angiography, or digital subtraction angiography) with stenosis of 50% or more in the artery feeding the acute ischemic territory.
   * Small vessel disease, defined by radiographic appearance consistent with ischemic infarction in the territory of a perforating arteriole, with ≤20 mm in diameter on axial sections and not involving the cortex, located in the white matter, internal or external capsule, deep brain nuclei, thalamus, or brainstem.
   * Evidence of a high-risk cardiac or aortic arch source of embolism (left ventricular or left atrial thrombus or "smoke," emboligenic valvular lesion or tumor, aortic arch plaque >3 mm thick or with mobile components or any other high-risk lesion)
   * Stroke of other determined cause such as presence of non-atherosclerotic vasculopathies (i.e. dissection, fibromuscular dysplasia), hypercoagulable states (must be tested in patients <55 years old) and hematologic disorders
2. Atrial septal defect or ventricular septal defect.
3. Coronary or valvular disease requiring surgical intervention.
4. Documented history of AF or atrial flutter.
5. Permanent indication for therapeutic oral anticoagulation at enrollment.
6. Already included in another clinical trial that will affect the objectives of this study.
7. Life expectancy <1 year.
8. Pregnancy.
9. Patient underwent or is scheduled for implantation of a pacemaker, implantable cardioverter defibrillator or cardiac resynchronization therapy device.
10. Unable or unwilling to follow the required procedures of the Clinical Investigation Plan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with a history of systemic embolization, i.e., cryptogenic stroke or acute peripheral arterial closures, and a concomitant PFO
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
incidence of first AF within 12 months after percutaneous PFO occlusion | 12 months
  to assess the incidence of first AF within 12 months after percutaneous PFO closure with a prespecified landmark analysis after 3 months to differentiate potentially device related AF (months 0-3) from likely intrinsic AF (months 4-12)

SECONDARY OUTCOMES:
Incidence of first AF within 3 months of continuous rhythm monitoring before the intended percutaneous PFO closure procedure | 3 months
  to assess the incidence of first AF within 3 months of continuous rhythm monitoring before PFo closure
Overall incidence of first AF from ICM-implantation to ICM-explantation or 36 months post implantation (if ICM remains in situ) excluding a blanking period of the first 3 months after PFO closure | 36 months
  To assess the overall incidence of first AF from ICM-implantation to ICM-explantation or 36 months post implantation
Differences in the primary endpoint according to the grade of the PFO | 12 months
  To assess the differences in the primary endpoint according to the grade of the PFO
Incidence of recurrent clinical embolic events such as cryptogenic strokes or systemic embolism including pulmonary embolism (with the use of the TOAST classification algorithm) | 36 months
  To assess the incidence of recurrent clinical embolic events
AF burden, defined as proportion of follow-up time with documented AF at different time points | 36 months
  To assess the AF burden
Incidence of major bleeding (BARC 3 to 5) | 36 months
  To assess the incidence of major bleeding
Incidence of any death and cardiovascular death at different timepoints | 36 months
  To assess the incicence of any death and cardiovascular death at diefferent timepoints
Device related events | 36 months
  To assess device related events

CONTACTS AND LOCATIONS:
Overall Officials: Raban Jeger, Prof Dr med, Principal Investigator — University Hospital, Basel, Switzerland; Tobias Reichlin, Prof Dr med, Principal Investigator — University Hospital Bern Inselspital, Switzerland
Locations (6):
- Switzerland (6):
  - Stadtspital Triemli, Zurich, Canton of Zurich
  - University Hospital Basel, Heart Center, Basel
  - University Hospital Bern Inselspital Cardiology, Bern
  - Cantonal Hospital St.Gallen Cardiology, Sankt Gallen
  - Bürgerspital Solothurn Cardiology, Solothurn
  - University Hospital Zürich Cardiology, Zurich

IPD SHARING:
Plan to Share IPD: No